CLINICAL TRIAL: NCT02476227
Title: Comparison of Operator-guided and Automatic Algorithm-guided Atrial Fibrillation Ablation. Randomized Open-labeled Study
Brief Title: Comparison of Operator-guided and Automatic Algorithm-guided Atrial Fibrillation Ablation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Military Institute od Medicine National Research Institute (Other)
Responsible Party: Principal Investigator, Marek Kiliszek, Principal Investigator, Military Institute od Medicine National Research Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1
Record Dates: First submitted 2015-06-05; First posted 2015-06-19 (Estimated); Last update posted 2018-03-29 (Actual); Status verified 2018-03

CONDITIONS: Atrial Fibrillation
Keywords: atrial fibrillation; pulmonary vein isolation; RF ablation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Visitag group (Experimental): Ablation using CARTO system. Visitag module: automated algorithm to collect RF ablation points using Visitag module. Criteria of ablation point: catheter stability range of motion ≤2.5mm, catheter stability time >15sec, contact force >5g over >50% of time. Optimal contact force suggested: 10-40g.
  Interventions: Procedure: Ablation using CARTO system
- Control group (Active Comparator): Ablation using CARTO system. Manual collection of RF ablation points by operator or by assistant. Optimal contact force suggested: 10-40g.
  Interventions: Procedure: Ablation using CARTO system

INTERVENTIONS:
Procedure: Ablation using CARTO system — automated algorithm (Visitag)-based vs. manual collection of RF ablation points during AF ablation
  Other Names: RF ablation (CARTO system); Pulmonary vein isolation (CARTO system)

SUMMARY:
Catheter ablation in the treatment of atrial fibrillation (i.e. pulmonary vein isolation) is now the most effective method of prevention of arrhythmia recurrence. Use of 3D electroanatomical system is now a golden standard.

Background hypothesis is that automatic algorithm collecting ablation points during pulmonary vein isolation (with certain catheter stability time, range of motion, and catheter-tissue contact force) prevents forming the gaps in the ablation line, thus preventing pulmonary vein reconnection and AF recurrence. The aim of the trial will be 1:1 comparison of the two methods of pulmonary vein isolation: with manual vs. automatic collection of ablation points using CARTO system and contact force catheter.

DETAILED DESCRIPTION:
Atrial fibrillation (AF) is the most common sustained supraventricular arrhythmia. It increases the risk of hospitalization and all-cause mortality. AF causes about 5-fold increase in the risk of stroke and 3-fold increase in the risk of heart failure.

Catheter ablation in the treatment of AF (i.e. pulmonary vein isolation) is now the most effective method of prevention of arrhythmia recurrence, especially in paroxysmal AF. Still, efficacy of one procedure in a 1-year follow-up is between 20 and 80%, depending on demographic and clinical factors (concomitant diseases), and on the form of the arrhythmia (paroxysmal-persistent), it also depends on the method of ablation used and the experience of the centre. In a big European registry including over 1,300 patients antiarrhythmic drugs-free efficacy of catheter ablation in AF in 1-year follow-up was about 40%. Major finding in patients with AF recurrence after catheter ablation is pulmonary vein reconnection, so decreasing the risk of pulmonary vein reconnections seems crucial to diminish the risk of AF recurrence. Several novel technologies have been proposed lately to improve efficacy of AF ablation, their real importance needs validation in a clinical trial.

Current standard is radiofrequency (RF) ablation with manual collection of ablation points (by operator or assistant). Automatic algorithm collect ablation points with additional criteria: catheter stability time, range of motion, and catheter-tissue contact force. The operator can see more precisely where the RF current has been applied and where are the gaps in the line.

Background hypothesis is that automatic algorithm collecting ablation points (with certain catheter stability time, range of motion, and catheter-tissue contact force) prevents forming the gaps in the ablation line, thus preventing pulmonary vein reconnection and AF recurrence. The aim of the trial will be 1:1 comparison of the two methods of pulmonary vein isolation: with manual vs. automatic collection of ablation points using CARTO system and contact force catheter.

ELIGIBILITY:
Inclusion Criteria:

* patients with symptomatic atrial fibrillation qualified to catheter ablation according to current standards

Exclusion Criteria:

* lack of informed consent
* two previous pulmonary vein isolations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2015-04; Primary Completion 2017-01 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
AF recurrence | 1-year follow-up after index procedure
  Number of AF recurrence after single catheter ablation during 12 months of follow-up.

SECONDARY OUTCOMES:
Arrhythmia-free survival | Time to arrhythmia recurrence, follow-up 3-18 months after index procedure
  Comparison of arrhythmia-free survival curves during the whole follow-up (even if extending over 1 year)

CONTACTS AND LOCATIONS:
Overall Officials: Marek Kiliszek, MD, PhD, Principal Investigator — Military Institute of Medicine
Locations (1):
- Military Institute of Medicine, Warsaw, Poland